CLINICAL TRIAL: NCT00725426
Title: A Study to Examine the Potential Effect of Rifampin on the Pharmacokinetics of Bosutinib When Administered Concomitantly to Healthy Subjects
Brief Title: Effect of Rifampin on Bosutinib When Both Are Given to Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3160A4-1106
Record Dates: First submitted 2008-07-24; First posted 2008-07-30 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: healthy subjects
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Bosutinib
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib

SUMMARY:
Study to examine whether rifampin has an effect on the pharmacokinetics of bosutinib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men age 18-50
* Healthy women of nonchildbearing potential, age 18-50

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (plasma concentrations) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Abbas R, Boni J, Sonnichsen D. Effect of rifampin on the pharmacokinetics of bosutinib, a dual Src/Abl tyrosine kinase inhibitor, when administered concomitantly to healthy subjects. Drug Metab Pers Ther. 2015 Mar;30(1):57-63. doi: 10.1515/dmdi-2014-0026. PMID 25803093